CLINICAL TRIAL: NCT02638883
Title: Implantation of the Cochlear™ Nucleus® Hybrid S Round Window (S-RW) in Adults
Status: Completed | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM 5630
Record Dates: First submitted 2015-12-03; First posted 2015-12-23 (Estimated); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Sensorineural Hearing Loss
Keywords: Adults; high frequency SNHL
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Implanted (Experimental): Subjects will be implanted with the Hybrid SRW cochlear implant.
  Interventions: Device: Hybrid SRW cochlear implant

INTERVENTIONS:
Device: Hybrid SRW cochlear implant — Subjects will be implanted with the Hybrid SRW

SUMMARY:
Evaluate the Cochlear™ Nucleus® S-Round Window (S-RW) implant in newly implanted adults with broader requirements to be considered an eligible candidate.

DETAILED DESCRIPTION:
The Food and Drug Administration recently approved the Cochlear Nucleus Hybrid L24 Implant System (P130016) for individuals aged 18 years and older who present with bilateral residual low frequency hearing sensitivity and severe to profound high frequency sensorineural hearing loss with limited benefit from appropriately fitted bilateral amplification. Additionally, the Nucleus Hybrid S12 Implant has been under evaluation since 2007 (IDE G#070016). The Nucleus Hybrid S-RW is a modification of the current Hybrid S12 implant. The Hybrid S-RW is designed to support implantation via a round window (RW) approach while maintaining the same relative insertion depth as the previous Hybrid S12 when implanted via cochleostomy

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older at the time of implantation
2. Sensorineural hearing loss with the following requirements: a pure tone threshold less (better) than or equal to 60 dB HL at 500 Hz,less than (better) or equal to 80 dB HL at 1500 Hz, and high frequency severe to profound (a threshold average of 2000, 3000, & 4000 Hz) of > 60dB HL.
3. Minimum of 30 days experience with appropriately fit bilateral amplification, fit as described in the Fitting and Use of Hearing Aids section below
4. Aided monosyllabic word score (e.g., CNC Word Test) (mean of two lists) between 20% and 60%, inclusive (i.e., 20% score 60%), in the ear to be implanted
5. Aided monosyllabic word score (e.g., CNC Word Test) (mean of two lists) in the contralateral ear equal to, or better than, the ear to be implanted but not more than 80%
6. Willingness to use bimodal stimulation (i.e., a cochlear implant on one ear and a hearing aid on the contralateral ear) through 12-months post-activation

Exclusion Criteria:

1. Individuals aged greater than 75 years
2. Duration of severe to profound hearing loss (above 2kHz) greater than 20 years
3. Medical or psychological conditions that contraindicate undergoing surgery as determined by the Investigator
4. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
5. Conductive overlay of 15 dB or greater at two or more frequencies, in the range 500 to 1000 Hz
6. Deafness due to lesions of the acoustic nerve or central auditory pathway
7. Active middle-ear infection or tympanic membrane perforation in the presence of active middle ear disease
8. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices as determined by the Investigator
9. Unwillingness or inability of the candidate to comply with all investigational requirements as determined by the Investigator
10. Additional handicaps that would prevent or restrict participation in the audiological evaluations as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Des Moines, Iowa, United States

REFERENCES:
- [Background] Gatehouse S, Noble W. The Speech, Spatial and Qualities of Hearing Scale (SSQ). Int J Audiol. 2004 Feb;43(2):85-99. doi: 10.1080/14992020400050014. PMID 15035561
- [Background] Noble W, Jensen NS, Naylor G, Bhullar N, Akeroyd MA. A short form of the Speech, Spatial and Qualities of Hearing scale suitable for clinical use: the SSQ12. Int J Audiol. 2013 Jun;52(6):409-12. doi: 10.3109/14992027.2013.781278. PMID 23651462
- [Background] PETERSON GE, LEHISTE I. Revised CNC lists for auditory tests. J Speech Hear Disord. 1962 Feb;27:62-70. doi: 10.1044/jshd.2701.62. No abstract available. PMID 14485785
- [Background] Spahr AJ, Dorman MF, Litvak LM, Van Wie S, Gifford RH, Loizou PC, Loiselle LM, Oakes T, Cook S. Development and validation of the AzBio sentence lists. Ear Hear. 2012 Jan-Feb;33(1):112-7. doi: 10.1097/AUD.0b013e31822c2549. PMID 21829134

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implanted
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Implanted
Number analyzed (Participants) | 6
Age, Customized [Count of Participants; unit: Participants] | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6
Age at Implant in Years [Mean (Standard Deviation); unit: years] | 57.5 (11.0)
Duration of Hearing Loss [Mean (Standard Deviation); unit: years] | 37.8 (25.2)

OUTCOME MEASURES:

1. Primary Outcome: CNC (Consonant-nucleus-consonant) Words
Description: Two CNC( consonant-nucleus-consonant) Word lists (Peterson & Lehiste, 1962) were administered in quiet at a level of 60 dBA in the sound-field and scored as a total number of words correct, expressed as a percentage. Possible score are range from 0% to 100 % words correctly repeated. Higher scores mean a better outcome.
Time Frame: 12 months
Population: Only 5 subjects were analysed rather than 6 as one subject used electric mode only by 12 months post activation.
Measure: Mean (Standard Deviation); unit: percentage of correct words.
Arm/Group | Implanted
Number analyzed (Participants) | 5
percentage of correct words. | 64.8 (23.0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Implanted
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted (N=6)
Sudden hearing threshold shift resulting in profound hearing loss (Ear and labyrinth disorders) | 1 (1)
Significant decrease in hearing thresholds (20-35dB) (Ear and labyrinth disorders) | 1 (1)
Skin Flap soreness (Skin and subcutaneous tissue disorders) | 1 (1) — Subject noticing some soreness at the magnet. Magnet strength was reduced from a 2 to 1. Still tender. Instructed patient to discontinue use until sore is fully healed
Open circuit electrodes (Product Issues) | 1 (1) — Resolved by deactivating the electrode.
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased tinnitus (Ear and labyrinth disorders) | 1 (1)
external otitis (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT02638883/Prot_000.pdf